CLINICAL TRIAL: NCT01656538
Title: A Randomized Phase II Study of Reolysin For Patients Receiving Standard Weekly Paclitaxel Therapy as Therapy For Advanced/Metastatic Breast Cancer
Brief Title: A Study of Reolysin For Patients With Advanced/Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I213
Record Dates: First submitted 2012-07-31; First posted 2012-08-03 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paclitaxel plus Reolysin (Experimental): Paclitaxel given weekly on days 1, 8, 15 every 4 weeks plus reolysin days 1, 2, 8, 9, 15 and 16.
  Interventions: Drug: Paclitaxel; Drug: Reolysin
- Paclitaxel (Active Comparator): Paclitaxel given weekly on days 1, 8 and 15 every 4 weeks.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel
Drug: Reolysin
  Arms: Paclitaxel plus Reolysin

SUMMARY:
Researchers doing this study want to evaluate the side effects of Reolysin when given together with paclitaxel. As these drugs have not been given together before, 6-9 patients will be treated with paclitaxel plus reolysin to ensure that side effects are tolerable.

DETAILED DESCRIPTION:
The purpose of the randomized part of this study is to find out if giving Reolysin in combination with paclitaxel can offer better results than standard therapy with paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological/cytological diagnosis of metastatic breast cancer.
* Patients must have advanced and/or metastatic disease, for which no curative therapy exists and for which systemic therapy is indicated.
* All patients must have an available formalin fixed paraffin embedded tissue block (from their primary or metastatic tumour) and must have provided informed consent for the release of the block, as well as for CTC and blood samples for correlative studies and banking.

For patients who have not had a tissue biopsy within the last 12 months, a repeat biopsy is strongly recommended but is not mandated providing that archival tissue is available.

• Re-biopsy is recommended if > 1 year since last biopsy.

* Presence of clinically and/or radiologically documented disease. All radiology studies must be performed within 28 days prior to randomization (within 35 days if negative).

All patients must have measurable disease as defined by RECIST 1.1.

The criteria for defining measurable disease are as follows:

Chest xray ≥ 20mm CT/MRI scan (with slice thickness <5mm) ≥10mm -> longest diameter Physical exam (using calipers) ≥ 10mm Lymph nodes by CT scan ≥ 15mm -> measured in short axis

* ECOG performance of 0, 1 or 2.
* Age ≥ 18 years of age

Previous Therapy

Surgery:

Previous major surgery is permitted provided that it has been at least 21days prior to patient randomization and that wound healing has occurred.

Chemotherapy:

Patients must have received at least one prior chemotherapy regimen for advanced or metastatic disease unless:

1. they have relapsed within 6 months of completion of adjuvant chemotherapy or
2. they have received taxane and/or anthracycline containing adjuvant chemotherapy.

Palliative therapy for breast cancer (chemotherapy, targeted, hormonal) is permitted but no more than three prior chemotherapy regimens are permissible.

Other Therapy:

Patients may have received other therapies including immunotherapy, or with signal transduction inhibitors.

Patients must have recovered from all reversible toxicity related to prior chemotherapy and have adequate washout from prior chemotherapy, and investigational agents as follows:

longest of one of the following.

* two weeks
* standard cycle length of prior regimen (i.e 21 days for doxorubicin q3 weeks)
* 5 half-lives for investigational drugs.

Radiation:

Prior external beam radiation is permitted provided a minimum of 4 weeks has elapsed between the last dose and enrollment to the trial. Exceptions may be made for low dose, non-myelosuppressive radiotherapy after consultation with NCIC CTG.

* Laboratory Requirements (must be done within 7 days prior to randomization)

Hematology:

Granulocytes (AGC) ≥ 1.5 x 10^9/L Platelets ≥ 100 x 10^9/L

Biochemistry:

* Serum creatinine ≤ 1.5 x ULN
* Total bilirubin ≤ 1.0 x ULN (unless elevated secondary to conditions such as Gilbert's disease)
* ALT and AST ≤ 3 x ULN (Note: ≤ 5 x ULN if documented liver metastasis)
* Proteinuria <2g/24hrs (screen using spot testing; if ≥ grade 2 repeat with mid-stream urine; if still ≥ grade 2, then urine collection for 24 hours to confirm <2g/24hrs).

Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.

Patients who cannot give informed consent (i.e. mentally incompetent patients, or those physically incapacitated such as comatose patients) are not to be recruited into the study. Patients competent but physically unable to sign the consent form may have the document signed by their nearest relative or legal guardian. Each patient will be provided with a full explanation of the study before consent is requested.

* Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 2 hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves that the patients registered on this trial will be available for complete documentation of the treatment, adverse events, response assessment and follow-up.
* In accordance with NCIC CTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies, except for adequately treated non-melanoma skin cancer or solid tumours curatively treated with no evidence of disease for ≥ 3 years. (Please call NCIC CTG if any questions about the interpretation of this criterion).
* Patients who are on immunosuppressive therapy or have known HIV infection or active hepatitis B or C.
* Patients with active or uncontrolled infections or with serious illnesses or medical conditions which would not permit the patient to be managed according to the protocol.
* Patients with significant cardiac (including uncontrolled hypertension) or pulmonary disease, or active CNS disease or infection.
* Patients are not eligible if they have a known hypersensitivity to the study drug(s) or their components.
* Patients with history of central nervous system metastases or untreated spinal cord compression.
* Patients who have contraindications to treatment with paclitaxel and/or neuropathy > grade 1.
* Women must be post-menopausal, surgically sterile or use two reliable forms of contraception while on study and for 6 months after discontinuing therapy. Women of childbearing potential must have a pregnancy test taken and proven negative within 7 days prior to randomization and must not be lactating. Men must be surgically sterile or use a barrier method of contraception.
* Concurrent treatment with other investigational drugs or anti-cancer therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-02-20 (Actual); Primary Completion 2016-11-18 (Actual); Study Completion 2018-02-14 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 24 months

SECONDARY OUTCOMES:
Response rate | 24 months
  To investigate additional potential measures of efficacy including Objective response rate, overall survival (OS) and CTC counts.
Tumour and tissue response of potential molecular factors | 24 months
  Potential molecular factors which may be prognostic or predictive of response by assessment of archival tumour tissue, CTCs, and serial blood samples
Number of patients with adverse events | 24 months
  To determine the tolerability and toxicity of reolysin and paclitaxel when given in combination.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Bernstein, Study Chair — BCCA - Vancouver Island Centre; Susan Ellard, Study Chair — BCCA-Cancer Ctr., Southern Interior
Locations (7):
- Canada (7):
  - BCCA - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Cancer Centre, Vancouver, British Columbia
  - BCCA - Vancouver Island Cancer Centre, Victoria, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bernstein V, Ellard SL, Dent SF, Tu D, Mates M, Dhesy-Thind SK, Panasci L, Gelmon KA, Salim M, Song X, Clemons M, Ksienski D, Verma S, Simmons C, Lui H, Chi K, Feilotter H, Hagerman LJ, Seymour L. A randomized phase II study of weekly paclitaxel with or without pelareorep in patients with metastatic breast cancer: final analysis of Canadian Cancer Trials Group IND.213. Breast Cancer Res Treat. 2018 Jan;167(2):485-493. doi: 10.1007/s10549-017-4538-4. Epub 2017 Oct 13. PMID 29027598